CLINICAL TRIAL: NCT03283241
Title: A Randomized, Multicentre, Double Blind, Parallel Study to Evaluate the Performance and Safety of the Zolidd One ExHex Dental Implant Compared to Uncoated One ExHex Dental Implant in Subjects With Partial Edentulism
Brief Title: Zolidd One ExHex Dental Implant Compared to Uncoated One ExHex Dental Implant in Subjects With Partial Edentulism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Addbio AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADD-001
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-01

CONDITIONS: Partial Edentulism

STUDY DESIGN:
Intervention Model Description: Parallel groups ration 1;1
Who Masked: Participant, Care Provider, Investigator
Masking Description: The devices are delivered single packed and sterile to distributor. The distributor performs blinding, randomization and distribution. The labels are, after blinding of lot number, identical for both the Active and the placebo device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zolidd One ExHex (Active Comparator): Coated titanium implant
  Interventions: Device: Zolidd One ExHex; Device: One ExHex
- One ExHex (Sham Comparator): Uncoated titanium implant
  Interventions: Device: Zolidd One ExHex; Device: One ExHex

INTERVENTIONS:
Device: Zolidd One ExHex — Subject will be treated/implanted at visit 2, one of the implants will be chosen as the "index implant"and will be followed together with other implants (maximum 6 implant per subject) at week 8,12 and month 12 and 24.
Device: One ExHex — Subject will be treated/implanted at visit 2, one of the implants will be chosen as the "index implant"and will be followed together with other implants (maximum 6 implant per subject) at week 8,12 and month 12 and 24.

SUMMARY:
A randomised, multicentre, double blind, parallel group comparative investigation where subjects will be randomised to receive coated or uncoated implants

DETAILED DESCRIPTION:
The study will consist of two parts. Part I, is the main study ending when all subjects have reached visit 5. The study will be evaluated and Clinical Study Report (CSR) will be written for this part.

Part II, of the study is a post-follow up study starting when the first subject has completed visit 5. There will be a separate CSR written for Study Part II.

The study Part I will begin with a baseline visit, visit 1, Informed consent procedure will take place. Provided the subject will give informed consent for both Study Part I and Study Part II the screening procedure starts. Subjects will undergo all screening and baseline assessment procedures including assessments of dental status to determine number of implants needed. Subjects who meet all the inclusion criteria and none of the exclusion criteria will be given a date for implant surgery within three weeks. The required number of implants will be ordered from the Study Distributor.

At the implantation day, visit 2, eligibility will be re-checked before the surgery procedures starts. The subjects who still are eligible will enter the treatment and the implantation surgery is conducted. The first follow-up visit after implantation will take place week 2 post-surgery and the last follow-up visit in Study Part I will be at week 12. Any post-surgical complications and adverse events will be collected and recorded in the eCRF. On demand, depending on the outcome of the surgery, additional visits might occur.

Study Part II, the Post Follow-up Study, consist of two visits, one at month 12 and another visit at month 24 post-surgery. Post-surgical complications and adverse events from Study Part I will be followed-up if not resolved previously. Safety, survival rate and marginal bone loss will be assessed and outcome recorded in the eCRF. Additional visits might occur depending on the status of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged >18 years
* Subjects should be willing to take part, able to understand the information given to them, and give written consent
* Subject diagnosed with partial edentulism and who needs at least one dental implant in the posterior upper jaw i.e. premolars to first molar. The same subject may also need implants in the posterior mandible (premolars to first molar region)

Exclusion Criteria:

* Suspected to be immunocompromised or are taking immunosuppressant
* Current participation in another clinical investigation or participation within the last 6 months
* Known sensitivity/allergies to any of the test materials or any of their ingredients, such as bisphosphonate, titanium or human fibrinogen
* Significant current or past medical history of hepatic, renal, cardiac, pulmonary, digestive, haematological, neurological, or psychiatric disease, hypercalcaemia, previous or ongoing malignancy in the head and neck region or uncontrolled diabetes type I which in the opinion of the Investigator, would compromise the safety of the subject or affect the outcome of the investigation
* Pregnant and lactating females or those actively seeking to become pregnant in the next 3 months
* Previous (last 5 years) or on-going Bisphosphonate or Denosumab treatment
* Significant marginal bone loss prior to implant insertion requiring bone grafting or bone graft substitute
* Subject with extraction(s) performed in the position of implant placement within the last 2 months
* Subject with need of >6 implants or a full bridge
* The final prosthetic construction in need of support from neighbouring teeth
* Known drug or alcohol abuse
* Subjects only needed implant(s) in the posterior mandible region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christer Dahlin, DDS, PhD, Principal Investigator — Käk kirurgiska kliniken NÄL, Trollhättan, Sweden
Locations (3):
- Sweden (3):
  - Dingletandläkarna, Dingle
  - Praktikertjänst AB Holmgatans Tandläkarmottagning, Falun
  - Käk-kirurgiska Kliniken, Näl, Trollhättan

IPD SHARING:
Plan to Share IPD: No
Not planned at the moment

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty two patient started the study
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | Zolidd One ExHex | One ExHex
Started | 32; 57 Implants | 30; 49 Implants
Completed 12 Weeks | 29; 50 Implants (Completed 12 weeks) | 29; 48 Implants (Completed 12 weeks)
Completed | 28; 44 Implants (Completed 24 month) | 27; 47 Implants (Completed 24 month)
Not Completed | 4; 13 Implants | 3; 2 Implants
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Subject relocated to Finland | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population Zolidd One exHex 32 One ExHex 30
Groups:
- Total: Total of all reporting groups
Arm/Group | Zolidd One ExHex | One ExHex | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (14.0) | 60.7 (12.4) | 58.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 16 | 15 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Stability at 12 Weeks Minus Value at Baseline (Day 1) Comparing Coated and Uncoated Implants Change in Stability From Day 1(Implantation to 12 Weeks After Implantation of the "Index Implant" Comparing Coated and Uncoated Implants
Description: The primary objective is to compare the mean change in stability at 12 weeks minus value at baseline (day 1)after surgery of the "index implant" between coated and uncoated implants.
  An ISQ (Implant Stability Quotient) probe is used to measure the stability of the implant ISQ (Implant Stability Quotient) scale is 1-100
  1 No stability 100 stability The aim is to get as close to a 100 as possible
Time Frame: 12 weeks
Population: At 12 weeks 3 subjects have missing data in Zolidd One ExHex and 1 subject have missing data in One ExHex
Measure: Mean (Standard Deviation); unit: ISQ (Implant Stability Quotient) score
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 29 | 29
ISQ (Implant Stability Quotient) score | 7.47 (25.71) | 2.83 (16.71)

2. Secondary Outcome: To Compare Absolute ISQ (Implant Stability Quotient) Highest Values Between Coated and Uncoated Implants for the "Index Implant" at Week 8 and Week 12
Description: To compare absolute ISQ (Implant Stability Quotient) highest values between coated and uncoated "index implants" at week 8 and week 12 after implantation An ISQ (Implant Stability Quotient) probe is used ISQ scale is 1-100
  1 No stability 100 stability Aim its to get close to 100
Time Frame: week 8 and week 12
Population: At 12 weeks 3 subjects have missing data in Zolidd One ExHex and 1 subject have missing data in One ExHex
Measure: Number; unit: ISQ Score
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 32 | 30
ISQ Score
  week 8 | 83 | 85
  week 12: number analyzed (Participants) | 29 | 29
  week 12 | 84 | 85

3. Secondary Outcome: Incidence of Post-surgery Complications and Adverse Events
Description: To compare safety as assessed by complications post-surgery and any other adverse event up to week 12 between all coated and all uncoated implants
Time Frame: Day1 to week 12
Population: This is the Adverse Event (AE) that has been reported and will be presented in the AE table under product issues, this is devices that failed and/or lossened At 12 weeks 3 subjects have missing data in Zolidd One ExHex and 1 subject have missing data in One ExHex
Measure: Number; unit: Number of events reported
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 29 | 29
Number of events reported | 5 | 4

4. Secondary Outcome: Change in ISQ (Implant Stability Quotient) Highest Value for the "Index Implant"
Description: To compare change in stability from day 1 to week 8 between the coated and the uncoated "index implants" An ISQ (Implant Stability Quotient) probe is used to measure the stability of the implant ISQ (Implant Stability Quotient) scale is 1-100
  1 No stability 100 stability The aim is to get as close to a 100 as possible
Time Frame: Day 1 to week 8
Population: In the Zolidd One ExHex 3 subjects have missing information. In the One ExHex group 1 subject have missing information at week 8 and 12.
Measure: Mean (Standard Deviation); unit: ISQ Score
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 29 | 29
ISQ Score | 4.34 (10.83) | 1.38 (8.86)

5. Secondary Outcome: Change in ISQ Highest Value for All Other Implants
Description: To compare change in stability from day 1 to week 8 and 12 between all other coated and all other uncoated implants An ISQ (Implant Stability Quotient) probe is used ISQ scale is 1-100
  1 No stability 100 stability
Time Frame: week 8 and week 12
Population: At 8 and 12 weeks 3 subjects have missing data in Zolidd One ExHex and 1 subject have missing data in One ExHex
Measure: Mean (Standard Deviation); unit: ISQ Score
Units Other Than Participants: Implants
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 29 | 29
Number analyzed (Implants) | 50 | 49
ISQ Score
  week 8 | 9.0 (21.6) | 5.1 (20.1)
  week 12: number analyzed (Implants) | 50 | 48
  week 12 | 7.1 (22.2) | 3.7 (20.4)

6. Secondary Outcome: Absolute ISQ (Implant Stability Quotient) Highest Value for All Other Implants
Description: To compare absolute ISQ (Implant Stability Quotient) highest value at week 8 and 12 between all other coated and all other uncoated implants An ISQ (Implant Stability Quotient) probe is used ISQ scale is 1-100
  1 No stability 100 stability
Time Frame: Week 8 and 12
Population: At 8 and 12 weeks 3 subjects have missing data in Zolidd One ExHex and 1 subject have missing data in One ExHex
Measure: Number; unit: ISQ Score
Units Other Than Participants: Implants
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 29 | 29
Number analyzed (Implants) | 50 | 49
ISQ Score
  week 8 | 83 | 85
  week 12: number analyzed (Implants) | 50 | 48
  week 12 | 84 | 85

7. Secondary Outcome: Change in Marginal Bone Height for All Other Implants
Description: To compare change in marginal bone height between all coated and all uncoated implants from at week 8 and 12 The marginal bone height is measured by x-ray and measuring the distance between the implant and bone in mm (millimeter)
Time Frame: week 8 and 12
Population: At 12 weeks 3 subjects have missing data in Zolidd One ExHex and 1 subject have missing data in One ExHex
Measure: Mean (Standard Deviation); unit: mm(milimeter)
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 29 | 29
mm(milimeter)
  Week 8 Mesial | 0.3 (0.7) | 0.2 (0.5)
  Week 8 Distal | 0.4 (0.8) | 0.2 (0.4)
  Week 12 Mesial | 0.5 (0.5) | 0.4 (0.7)
  Week 12 Distal | 0.6 (1.0) | 0.4 (0.6)

8. Secondary Outcome: Post-surgical Complications and Other Adverse Events (AEs) for All Implants
Description: To compare safety as assessed by complications post-surgery and other adverse events up to month 24 post-implantation visit between all coated and all uncoated implants
Time Frame: month 24
Population: See adverse events, all implant loss is reported as adverse events
Measure: Number; unit: Number of events reported
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 32 | 30
Number of events reported | 4 | 1

9. Secondary Outcome: Survival Rate for All Implants
Description: To compare survival rate of implants up to 24 months between all coated and all uncoated implants
Time Frame: 24 months
Population: At 24 month 4 subjects have missing data in Zolidd One ExHex (28 subjects) and 3 subjects have missing data in One ExHex (27 subjects)
Measure: Mean (95% Confidence Interval); unit: Number of implant loss
Units Other Than Participants: Implants
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 28 | 27
Number analyzed (Implants) | 44 | 47
Number of implant loss | 0.930 [0.824 to 0.973] | 0.939 [0.822 to 0.980]

10. Secondary Outcome: Change in Marginal Bone Height for All Implants
Description: To compare change in marginal bone height from day 1 to month 12 and 24 between all coated and all uncoated implants The marginal bone height is measured by x-ray and measuring the distance between the implant and bone in mm (millimeter)
Time Frame: Day 1, month 12 and 24
Population: At 12 weeks 3 subjects have missing data in Zolidd One ExHex (29 subjects) and 1 subject have missing data in One ExHex (29 subjects) At 24 month 4 subjects have missing data in Zolidd One ExHex (28 subjects) and 3 subjects have missing data in One ExHex (27 subjects)
Measure: Mean (Standard Deviation); unit: mm(millimeter)
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 32 | 30
mm(millimeter)
  Week 12 Mesial: number analyzed (Participants) | 29 | 29
  Week 12 Mesial | 0.5 (0.8) | 0.3 (0.6)
  Week 12 Distal: number analyzed (Participants) | 29 | 29
  Week 12 Distal | 0.5 (0.9) | 0.3 (0.6)
  Month 24 Mesial: number analyzed (Participants) | 28 | 27
  Month 24 Mesial | 0.5 (1.0) | 0.5 (1.0)
  Month 24 Distal: number analyzed (Participants) | 28 | 27
  Month 24 Distal | 0.5 (1.0) | 0.5 (1.0)

11. Secondary Outcome: Occurrence of Signs Associated With Peri-implantitis for All Implants
Description: To compare peri-implantitis frequency at 12 and 24 months between all coated and all uncoated implants Ocular assessment of redness and swelling this is an overall judgement of peri-implantitis
Time Frame: Month 12 and 24
Population: At 12 and 24 month 4 subjects have missing data in Zolidd One ExHex (28 subjects) and 3 subjects have missing data in One ExHex (27 subjects)
Measure: Number; unit: number of participants redness/swollen
Arm/Group | Zolidd One ExHex | One ExHex
Number analyzed (Participants) | 32 | 30
number of participants redness/swollen
  12 month: number analyzed (Participants) | 28 | 27
  12 month | 0 | 0
  24 month: number analyzed (Participants) | 28 | 27
  24 month | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected from visit 1 to 24 month
Arm/Group | Zolidd One ExHex | One ExHex
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/30
Other Adverse Events (participants affected / at risk) | 7/32 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolidd One ExHex (N=32) | One ExHex (N=30)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolidd One ExHex (N=32) | One ExHex (N=30)
Device Failure (Product Issues) | 7 (9) | 4 (4)
Back pan (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03283241/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT03283241/SAP_001.pdf